CLINICAL TRIAL: NCT01429948
Title: Novel Biomarkers for Personalized Therapy in Korean Patients With Ischemic Stroke
Brief Title: Identification the Cause of Silent Cerebral infarctiON in Healthy Subjects (ICONS)
Acronym: ICONS
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-02-046
Record Dates: First submitted 2011-09-06; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Cerebral Infarction
Keywords: Stroke, Ischemic; Patent foramen ovale; Magnetic resonance imaging; Paradoxical embolism; Transcranial Doppler; Silent cerebral infarct
MeSH Terms: conditions — Cerebral Infarction; Ischemic Stroke; Foramen Ovale, Patent; Embolism, Paradoxical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Case group: Healthy subjects with silent cerebral infarction
- Control group 1: Patients with acute cryptogenic embolic stroke
- Control group 2: Patients with acute stroke with conventional stroke mechanisms

SUMMARY:
We hypothesized that paradoxical embolism may be one of the main mechanisms of silent cerebral infarction (SCI) located outside the perforating artery territory. In the present study, we evaluated the association between SCI and paradoxical embolism detected by agitated saline transcranial Doppler (TCD) monitoring in healthy subjects without history of stroke or transient ischemic attack (TIA). We also compared the frequency and amount of paradoxical embolism between healthy subjects with SCI and acute stroke patients with presumed cryptogenic embolism or conventional stroke mechanisms.

ELIGIBILITY:
Inclusion Criteria:

Healthy subjects

* Subjects with age over 20 years
* Subjects who consecutively visited a health promotion center for a health screening examination that included routine laboratory test, cardiac work-ups (12-lead electrocardiography and/or echocardiography), and brain magnetic resonance image (MRI) and MR angiography (MRA)
* Subjects who showed silent brain infarction (SCI) which was defined as a focal hyperintensity lesion 3 mm or large in diameter in the fluid-attenuation inversion recovery (FLAIR) images without a history of a corresponding stroke or transient ischemic attack (TIA)
* Subjects who performed agitated saline transcranial Doppler (TCD) monitoring

Patients with acute stroke (both cryptogenic embolic stroke and conventional stroke mechanisms)

* Patients with age over 20 year
* Patients with focal neurologic deficits presented within 7 days of symptom onset
* Patients with acute ischemic lesions on diffusion-weighted image (DWI)
* Patients who performed agitated saline TCD monitoring

Exclusion Criteria:

Healthy subjects

* Subjects with the presence of previous history of stroke or TIA
* Subjects with the presence of dementia on history taking or mini-mental status examination
* Subjects with the presence of proximal source of embolism, including atrial fibrillation or significant (≥50%) stenosis on cervicocerebral artery on MRA or carotid Duplex
* Subjects who had SCI restricted within perforator territory (basal ganglia or pons) suggesting that microangiopathy rather than embolism could be the main mechanism of SCI
* Subjects in whom agitated saline TCD monitoring was not performed or those who had poor temporal windows

Patients with acute stroke (both cryptogenic embolic stroke and conventional stroke mechanisms)

* Patients in whom agitated saline TCD monitoring was not performed or those who had poor temporal windows

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Hospital
Sampling Method: Probability Sample
Enrollment: 581 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Frequency and amount of right-to-left shunts (RLS) on agitated saline TCD monitoring | Within a month after MRI scanning

CONTACTS AND LOCATIONS:
Overall Officials: Oh Young Bang, MD, PhD, Principal Investigator — Samsung Medical Center, Sungkyunkwan University
Locations (1):
- Samsung Medical Center, Sungkyunkwan University, Seoul, South Korea

REFERENCES:
- [Derived] Kim SJ, Shin HY, Ha YS, Kim JW, Kang KW, Na DL, Bang OY. Paradoxical embolism as a cause of silent brain infarctions in healthy subjects: the ICONS study (Identification of the Cause of Silent Cerebral Infarction in Healthy Subjects). Eur J Neurol. 2013 Feb;20(2):353-60. doi: 10.1111/j.1468-1331.2012.03864.x. Epub 2012 Sep 9. PMID 22958084